CLINICAL TRIAL: NCT01839383
Title: The Effects of Different Dialysate Calcium Concentration on Mineral-bone Metabolism in Chinese Patients on Maintenance Hemodialysis
Brief Title: The Effects of Different Dialysate Calcium Concentration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJFH-EC/2013-020
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Mineral-bone Metabolism

ARMS (3):
- DCa1.25 (Active Comparator): using dialysate calcium concentration 1.25 mmol/L(DCa1.25)
  Interventions: Other: different dialysate calcium concentration
- DCa1.5 (Active Comparator): using dialysate calcium concentration 1.5mmol/L
  Interventions: Other: different dialysate calcium concentration
- DCa1.75 (Active Comparator): using dialysate calcium concentration 1.75mmol/L
  Interventions: Other: different dialysate calcium concentration

INTERVENTIONS:
Other: different dialysate calcium concentration

SUMMARY:
The investigators enrolled 90 patients on maintenance hemodialysis with dialytic vintage ≥12 months, iPTH 150-300pg/ml and serum calcium<2.5mmol/L. Patients were randomized to three groups with different dialysate calcium concentration , 1.25 mmol/L(DCa1.25), 1.5mmol/L(DCa1.5) and 1.75 mmol/L(DCa1.75) for 24 months respectively. Hemodialysis was performed for 4 hours three times weekly. Serum total calcium(tCa), ionized calcium(iCa),intact parathyroid hormone(iPTH)and phosphorus (P) levels were recorded before and after the study and single dialysis session in every patient. iCa and P levels were measured in spent dialysate.Bone density, bone-specific alkaline phosphatase(BAP), osteoprotegerin(OPG)、β-crosslaps、total Procollagen Type I Intact Propeptide (P1NP）and vascular calcification were measured in every patient periodically. vascular calcification including aortic arch calcification, abdominal aorta calcification and coronary artery calcification were measured by chest radiography, lateral lumbar radiographs and coronary artery computer tomography (CT) respectively. The primary endpoints included death, cardio-cerebral vascular disease(defined as heart failure, myocardial infarction and stroke), newly nontraumatic bone fracture, secondary parathyroidism uncontrolled by medicine and valvular or vascular calcification. The secondary endpoint were admission or emergency observation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, maintenance hemodialysis, dialytic vintage ≥12 months, iPTH 150-300pg/ml, serum calcium<2.5mmol/L, serum calcium<2.5mmol/L.

Exclusion Criteria:

* Age<18 or >65 Severe acid-base disturbance History of parathyroid glands or adrenal gland combined with consumptions or malnutrition anemia due to acute bleeding or other diseases except for renal failure newly occurred bone fracture within 3 months active stage of immunological diseases using glucocorticoid or immunosuppressor combined with any disease with expect duration <2 year newly occurred acute heart failure, acute myocardial failure , acute cerebral infarction or stroke within 6 months pregnant women of women in preparation for pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
death | 24months
  incidence of death
cardio-cerebral vascular disease(defined as heart failure, myocardial infarction and stroke) | 24months
  incidence of cardio-cerebral vascular disease
newly nontraumatic bone fracture | 24months
  incidence of newly nontraumatic bone fracture
secondary hyperparathyroidism uncontrolled by medicine | 24months
  incidence of secondary hyperparathyroidism uncontrolled by medicine
valvular or vascular calcification | 24months
  incidence of valvular or vascular calcification

SECONDARY OUTCOMES:
admission or emergency observation | 24months
  incidence of admission or emergency observation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship hospital, Beijing, Beijing Municipality, China